CLINICAL TRIAL: NCT01409408
Title: Comparison Between Amlodipine and Aliskiren in Diabetic Hypertensive Patient With Blood Pressure Not Controlled by Losartan: Effects on Endothelial Function and Renin Concentration and Activity
Brief Title: Comparison of Amlodipine and Aliskiren in Diabetic Hypertensive Patient With Blood Pressure Not Controlled by Losartan
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to preliminary results of Altitude Trial.
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Collaborators: Novartis (Industry)
Responsible Party: Ronaldo Altenburg Odebrecht Curi Gismondi, Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAALIDH
Record Dates: First submitted 2011-08-01; First posted 2011-08-04 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension; Diabetes Mellitus
Keywords: Hypertension; Diabetes Mellitus; Vascular stiffness; Endothelial function
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Active Comparator)
  Interventions: Drug: Aliskiren
- Amlodipine (Active Comparator)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Aliskiren — 300 mg of aliskiren daily for 8 weeks.
  Other Names: Rasilez.
  Arms: Aliskiren
Drug: Amlodipine — Amlodipine 5 mg daily for 8 weeks.
  Other Names: Norvasc.
  Arms: Amlodipine

SUMMARY:
Assess if aliskiren is capable of enhancing vascular stiffness and endothelial function and compare theses effects and renin activity and concentration to those obtained with a calcium channel blocker, amlodipine, in patients with diabetes mellitus type 2 and blood pressure not controlled by 100 mg per day of losartan.

DETAILED DESCRIPTION:
Hypertension and diabetes mellitus are important risk factors for cardiovascular morbidity and mortality. Endothelial dysfunction and vascular rigidity are two pathophysiological mechanisms that may explain this relationship. Recent publications showed that both ACEi (angiotensin converting enzyme inhibitor) and ARB (angiotensin receptor blocker) were capable of improving vascular stiffness and endothelial function, and that these effects occurred despite blood pressure reduction. The major debate that persists is which drug to associate with ACEi or ARB to achieve blood pressure control in diabetic patients. Recent studies showed that even in patients under ACEi or ARB therapy there may be residual activity in the renin-angiotensin-aldosterone system (RASS). Direct renin inhibitors (DRI) are a new class of anti-hypertensive drugs that may complement the blockade of the RASS. Aliskiren was the first drug of this class that completed phase 3 studies and marketed in the 21th century. It's main advantage is that DRI may reduce angiotensin II and aldosterone synthesis without increasing renin levels. This study main objective is to assess if aliskiren is capable of enhancing vascular stiffness and endothelial function and compare theses effects to those obtained with a calcium channel blocker, amlodipine, in patients with diabetes mellitus type 2 and blood pressure not controlled by 100 mg per day of losartan. Vascular stiffness and endothelial function will be measured by: pulse wave velocity, augmentation index, brachial artery flow-mediated vasodilation, peripheral arterial tonometry (EndoPat). Another main objective is to compare plasma renin activity and concentration between those groups.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatorial patients with age between 40 and 70 years-old.
* Systemic arterial hypertension previously diagnosed and in use of two or less anti-hypertensive drugs in the preceding 4 weeks.
* Those patients without anti-hypertensive drug prescribed in the last 4 weeks with office systolic blood pressure between 140 and 159 mmHg and diastolic between 90 and 109 mmHg.
* Type 2 diabetes mellitus in use of oral medication that were not changed in the preceding 4 weeks. Glycated hemoglobin A1c less than 9.0%.
* Accepted the consent form.

Exclusion Criteria:

* Office systolic blood pressure equal or more than 180 mmHg, with or without treatment
* Office diastolic blood pressure equal or more than 110 mmHg, with or without treatment
* Evidences of a secondary cause for hypertension
* Glycated hemoglobin A1c > 9.0%
* Insulin therapy
* Chronic kidney disease of level 3 to 5 or in dialysis
* Advanced target organ lesion, obtained by history or additional exams, and defined by: previous myocardial infarction, heart failure with ejection fraction less than 40%, cerebral vascular accident (ischemic or hemorrhagic), peripheral vascular disease (claudication or doppler with obstruction > 50% of vascular lumen), retinopathy with visual loss, symptomatic neuropathy.
* Cardiac arrhythmias, except for ectopic beats
* Any clinical or disabling condition that, in the opinion of the investigators, may confound or prejudice study results.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Vascular stiffness | 8 weeks
  Vascular stiffness will be measured by pulse wave velocity and augmentation index and compared between anlodipine and aliskiren.
Endothelial function | 8 weeks
  Access endothelial function by peripheral arterial tonometry and brachial flow-mediated vasodilation and compare it between anlodipine and aliskiren.
Renin activity and concentration | 8 weeks
  Access plasma renin activity and concentration and compare it between anlodipine and aliskiren.

SECONDARY OUTCOMES:
Compare drug effects in office blood pressure measurements to those obtained by home blood pressure monitoring and ambulatory blood pressure monitoring | 8 weeks
  Compare drug effects in office blood pressure measurements to those obtained by home blood pressure monitoring and ambulatory blood pressure monitoring
Assess drugs effects in renin-angiotensin-aldosterone system (RAAS) and correlate it to renin concentration/mass and plasmatic renin activity | 8 weeks
  Assess drugs effects in RAAS and correlate it to renin concentration/mass and plasmatic renin activity
Correlation of drug effects and uric acid plasmatic concentration | 8 weeks
  Correlation of drug effects and uric acid plasmatic concentration
Correlation of drug effects and glomerular filtration rate | 8 weeks
  Correlation of drug effects and glomerular filtration rate
Correlation of drug effects and microalbuminuria | 8 weeks
  Correlation of drug effects and microalbuminuria
Correlation of drug effects and left ventricular mass and function (systolic and diastolic) | 8 weeks
  Correlation of drug effects and left ventricular mass and function (systolic and diastolic)

CONTACTS AND LOCATIONS:
Overall Officials: Ronaldo A Gismondi, MD, DsC, Principal Investigator — HUPedroernesto (UERJ); Mario F Neves, MD, PhD, Study Director — HUPedroernesto (UERJ); Wille Oigman, MD, PhD, Study Chair — HUPedroernesto (UERJ)
Locations (1):
- Hospital Universitario Pedro Ernesto, Rio de Janeiro, Rio de Janeiro, Brazil